CLINICAL TRIAL: NCT03818126
Title: The Del Nido Cardioplegia Versus the Cold Blood Cardioplegia in Adult Patients Undergoing Aortic Valve Replacement
Brief Title: The Del Nido Versus Cold Blood Cardioplegia in Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pawel Buszman (Other)
Responsible Party: Sponsor-Investigator, Pawel Buszman, Chief Executive Officer, American Heart of Poland
Organization: American Heart of Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DELNIDO01
Record Dates: First submitted 2019-01-20; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Aortic Valve Disease; Ischemia-reperfusion Injury
Keywords: del Nido; cardioplegia; aortic valve
MeSH Terms: conditions — Aortic Valve Disease; Reperfusion Injury | interventions — Del Nido cardioplegia solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- del Nido cardioplegia (Experimental)
  Interventions: Drug: del Nido cardioplegia
- cold blood cardioplegia (Active Comparator)
  Interventions: Drug: cold blood cardioplegia

INTERVENTIONS:
Drug: del Nido cardioplegia — The del Nido components are: Plasma-Lyte A (1000ml), Mannitol 20% (16.3ml), MgSO4 50% (4ml) , NaHCO3 8.4% (13ml) , KCl 2mEq/mL (13ml), Lidocaine 1% (13ml). This solution is mixed with autologous patient blood from the cardiopulmonary circuit in a 4:1 ratio (crystalloid:blood).
  The dosage is 20ml/kg. The target administration pressure is 100-200mmHg and the target administration flow is 200-300ml/min. The solution temperature is 4 degrees Celsius. Additional dose of the cardioplegia is given only if the cross-clamp time exceeds 90 minutes. Due to high volume given in a single delivery, 40 milligrams of furosemide are injected into cardiopulmonary circuit.
  Arms: del Nido cardioplegia
Drug: cold blood cardioplegia — The cold blood cardioplegia components are: Plasma-Lyte A (435ml), Mannitol 15% (20ml), NaHCO3 8.4% (20ml), KCl 2mEq/mL (25ml). The solution is mixed with autologous patient blood from the cardiopulmonary circuit in a 1:4 ratio (crystalloid:blood).
  The initial dose is 15ml/kg and a dose of 5ml/kg is added every 20-30 minutes or whenever cardiac activity is observed. The target administration pressure is 100-200mmHg and the target administration flow is 200-300ml/min. The solution temperature is 4 degrees Celsius.
  Arms: cold blood cardioplegia

SUMMARY:
A group of 150 patients undergoing aortic valve replacement procedure will be randomized either into del Nido cardioprotection protocol (75 participants) or into the cold blood cardioplegia protocol (75 participants).

The intraoperative and perioperative outcomes of using each solution will be presented and compared (see the endpoints).

DETAILED DESCRIPTION:
The del Nido cardioplegia was developed by Pedro del Nido and his team at the University of Pittsburgh in 1990s. It was primarily designed for children and it has been used in pediatric cardiac surgery in Boston's Children Hospital since 1994.

There are few studies regarding the del Nido cardioplegia. A prospective, randomized trial was designed to determine the efficiency of the del Nido cardioplegia when compared to multidose cold blood cardioplegia in cardiac procedures with short and moderate cross-clamp times.

For the analysis of two cardioprotection protocols, it is essential to compare groups equal in terms of the surgery and perioperative care, with the same surgical risk and cross-clamp time. The research required elimination of all the unnecessary variables.

The patients undergoing aortic valve replacement procedure were selected as a study population. A group of 150 patients will be randomized either into del Nido cardioprotection protocol (75 participants) or into the cold blood cardioplegia protocol (75 participants).

The intraoperative and perioperative outcomes of using each solution will be presented and compared (see the endpoints).

ELIGIBILITY:
Inclusion Criteria:

* qualification for isolated aortic valve replacement
* age>18 years
* given consent for the study

Exclusion Criteria:

* reoperation
* allergy to lidocaine
* coronary artery disease requiring surgical or percutaneous intervention
* pregnancy
* ejection fraction<30%
* massive aortic calcification ("porcelain aorta")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Electrical cardiac activity during cross-clamp | intraoperative
  Electrical activity observed during the cardiac arrest (cross-clamp)
Ventricular fibrillation during reperfusion | intraoperative
  Ventricular fibrillation as first observed rhythm after removing the aortic cross-clamp
hs-TnT (High sensitivity troponin T) - 24 hours | 24 hours postoperatively
  High sensitivity troponin T measured 24 hours postoperatively
hs-TnT (High sensitivity troponin T) - 48 hours | 48 hours postoperatively
  High sensitivity troponin T measured 48 hours postoperatively
CK-MB (Creatine kinase- MB isoenzyme) - 24 hours | 24 hours postoperatively
  Creatine kinase (MB isoenzyme) measured 24 hours postoperatively
CK-MB (Creatine kinase- MB isoenzyme) - 48 hours | 48 hours postoperatively
  Creatine kinase (MB isoenzyme) measured 48 hours postoperatively

SECONDARY OUTCOMES:
Ventricular fibrillation during the cardioplegia administration | intraoperative
Time from the beginning of cardioplegia administration to cardiac arrest | intraoperative
Procedural use of the pacemaker | intraoperative
Intraoperative myocardial infarction | intraoperative
Fall of ejection fraction (EF) | 48 hours
  5% fall in the EF
Inotrope administration | intraoperative, 48 hours
Use of the intraaortic balloon pump | intraoperative, 48 hours
Perioperative atrial fibrillation | up to 2 weeks
Perioperative arrhythmia (other than AF) | up to 2 weeks
Postoperative packed red blood cells transfusion | up to 2 weeks
Perioperative creatinine values | up to 2 weeks
Kidney injury | up to 2 weeks
  The creatinine elevation >25% or >0.5mg/dl
CVVHDF | up to 2 weeks
  Use of continous veno-venous hemodiafiltration
Cardiac death | 30 days postoperative
  death from cardiac reasons (e.g. myocardial infarction, low ejection fraction, arrhythmia).
Overall mortality | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Marek Cisowski, MD,PhD, Principal Investigator — 1st Department of Cardiac Surgery, American Heart of Poland, Bielsko-Biala, Poland
Locations (1):
- 1st Department of Cardiac Surgery, Bielsko-Biala, Poland

IPD SHARING:
Plan to Share IPD: No